CLINICAL TRIAL: NCT01918033
Title: A Phase III, Multi-Center, Randomized, Parallel-Group, Placebo-Controlled and Double- Blind Trial to Study the Efficacy and Safety of MK-4117 in Japanese Subjects With Perennial Allergic Rhinitis
Brief Title: A Study of the Efficacy and Safety of Desloratadine (MK-4117) in Japanese Participants With Perennial Allergic Rhinitis (MK-4117-200)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4117-200; 132244 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Rhinitis; Allergic Rhinitis; Nose Diseases; Respiratory Tract Diseases; Immune System Diseases; Cholinergic Antagonists; Cholinergic Agents; Neurotransmitter Agents; Histamine H1 Antagonists, Non-Sedating; Histamine H1 Antagonists; Histamine Antagonists; Histamine Agents
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis; Rhinitis, Allergic; Nose Diseases; Respiratory Tract Diseases; Immune System Diseases | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desloratadine 5 mg (Experimental): Participants receive one desloratadine 5 mg tablet and one placebo tablet orally once daily for up to 2 weeks
  Interventions: Drug: Desloratadine 5 mg; Drug: Placebo
- Desloratadine 10 mg (Experimental): Participants receive two desloratadine 5 mg tablets orally once daily for up to 2 weeks
  Interventions: Drug: Desloratadine 5 mg
- Placebo (Placebo Comparator): Participants receive two placebo tablets orally once daily for up to 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desloratadine 5 mg — Desloratadine 5 mg tablets
  Arms: Desloratadine 10 mg; Desloratadine 5 mg
Drug: Placebo — Matching placebo to desloratadine 5 mg tablets
  Arms: Desloratadine 5 mg; Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of desloratadine (MK-4117) in Japanese participants with perennial allergic rhinitis. The primary hypothesis is that desloratadine is superior to placebo after 2 weeks of treatment with regard to change from baseline in Total Nasal Symptom Score among Japanese participants with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with perennial allergic rhinitis
* Outpatient.

Exclusion Criteria:

* Lower respiratory tract infection or nasopharyngolaryngeal infection (acute upper respiratory tract infection, acute pharyngolaryngitis, or acute tonsillitis, etc.)
* Coexisting infections or systemic mycosis for which there are no effective antibiotics
* Asthma complication under treatment
* Nasal septum ulcers, nasal surgery, or nasal trauma, which has not healed
* Vasomotor rhinitis or eosinophilic rhinitis
* Nasal conditions (infectious sinusitis, hypertrophic rhinitis, acute or chronic rhinitis, nasal polyps, septal deviation, etc.) which may interfere with the evaluation of the efficacy of the study drug
* History of hypersensitivity to antihistamines or study drug
* Currently receiving treatment with another investigational drug or has received an investigational drug in the past 3 months
* Has started specific desensitization therapy or nonspecific allassotherapy (Histaglobin, vaccine therapy, etc.) or who had discontinued such therapies within 90 days (3 months) before the day of obtaining informed consent
* Severe hepatic, renal, cardiac, hematological disease, or other serious coexisting diseases and whose general condition is poor
* History of malignancy or clinically important hematological disorder
* History of severe drug allergy (e.g., anaphylactoid reaction).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2014-01-26 (Actual); Study Completion 2014-01-26 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okamoto Y, Maeda Y, Oshima N, Hisada S. A Phase III clinical trial of desloratadine in Japanese subjects with perennial allergic rhinitis: A randomized controlled trial. J Clin Therapeut Med. 2016;32(12):967-978 [in Japanese] https://mol.medicalonline.jp/archive/search?jo=an9cltmd&ye=2016&vo=32&issue=12

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Started | 203 | 203 | 202
Treated | 202 (One randomized participant did not receive study drug.) | 203 | 201 (One randomized participant did not receive study drug.)
Completed | 198 | 201 | 199
Not Completed | 5 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo | Total
Number analyzed (Participants) | 203 | 203 | 202 | 608
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (13.1) | 33.7 (11.9) | 34.7 (12.6) | 34.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 105 | 121 | 342
  Male | 87 | 98 | 81 | 266

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Assessed by the Investigator at Week 2
Description: The investigator interviewed and examined participants to evaluate for nasal symptoms of: sneezing (daily frequency of attacks; score of 0=less than 1 time to 3=11+ times), rhinorrhea (daily frequency of blowing nose; score of 0=less than 1 time to 3=11+ times), nasal congestion (score of 0=less than nasal blockage without oral breathing to 3=severe nasal blockage causing prolonged oral breathing in a day), and nasal itching (score of 0=none to 3=nose is itchy, requiring frequent rubbing or blowing nose). The TNSS is the sum of the 4 nasal symptom sub-scores. TNSS scores could range from 0 to 12, with a higher score indicating more frequent/severe nasal symptoms.
Time Frame: Baseline and Week 2
Population: The Full Analysis Set (FAS) population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for TNSS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale | -1.96 (2.21) [-2.25 to -1.67] | -1.94 (2.21) [-2.23 to -1.65] | -1.87 (2.34) [-2.16 to -1.58]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.661, Constrained Longitudinal Data Analysis; Model with terms for visit, visit-by-treatment, visit-by-age strata, visit-by-severity interactions; visit treated as a categorical variable; Difference in Least Squares (LS) Means = -0.09, 95% CI 2-sided [-0.49 to 0.31] — Difference in LS Means for Change from Baseline in TNSS at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.707, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.08, 95% CI 2-sided [-0.48 to 0.32] — Difference in LS Means for Change from Baseline in TNSS at Week 2

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE is defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of the study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug, is also an AE. The number of participants who experienced an AE, regardless of causality or severity, was summarized.
Time Frame: Up to Week 4
Population: The All-Subjects-as-Treated (ASaT) population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Participants | 27 | 29 | 20

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE
Description: An AE is defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of the study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug, is also an AE. The number of participants who discontinued study drug, whether permanently or temporarily, due to an AE was summarized.
Time Frame: Up to Week 2
Population: The ASaT population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Participants | 1 | 0 | 2

4. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Assessed by the Investigator at Day 3 and Week 1
Description: as for outcome 1
Time Frame: Baseline and Day 3, Week 1
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for TNSS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Change from Baseline (BL) at Day 3 | -1.12 (2.05) [-1.38 to -0.86] | -1.11 (2.02) [-1.37 to -0.85] | -0.63 (2.03) [-0.89 to -0.37]
  Change from BL at Week 1 | -1.39 (2.41) [-1.68 to -1.09] | -1.39 (2.28) [-1.69 to -1.10] | -1.48 (2.32) [-1.78 to -1.18]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.010, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.48, 95% CI 2-sided [-0.84 to -0.11] — Difference in LS Means for Change from Baseline in TNSS at Day 3
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.013, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.46, 95% CI 2-sided [-0.82 to -0.10] — Difference in LS Means for Change from Baseline in TNSS at Day 3
Statistical Analysis 3: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.569, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.12, 95% CI 2-sided [-0.29 to 0.53] — Difference in LS Means for Change from Baseline in TNSS at Week 1
Statistical Analysis 4: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.685, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.09, 95% CI 2-sided [-0.33 to 0.50] — Difference in LS Means for Change from Baseline in TNSS at Week 1

5. Secondary Outcome: Change From Baseline in Nasal Symptom Sub-Scores Assessed by the Investigator
Description: The investigator interviewed and examined participants to evaluate for nasal symptoms of: sneezing (daily frequency of attackes; score of 0=less than 1 time to 3=11+ times), rhinorrhea (daily frequency of blowing nose; score of 0=less than 1 time to 3=11+ times), nasal congestion (score of 0=less than nasal blockage without oral breathing to 3=severe nasal blockage causing prolonged oral breathing in a day), and nasal itching (score of 0=none to 3=nose is itchy, requiring frequent rubbing or blowing nose). Nasal symptom sub-scores could range from 0 to 3, with a higher nasal symptom sub-score indicating more frequent/severe nasal symptoms.
Time Frame: Baseline and Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for nasal symptom sub-scores as assessed by the investigator.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Sneezing: Change from BL at Day 3 | -0.21 (0.75) [-0.30 to -0.13] | -0.29 (0.67) [-0.38 to -0.20] | -0.13 (0.65) [-0.21 to -0.04]
  Sneezing: Change from BL at Week 1 | -0.27 (0.78) [-0.36 to -0.17] | -0.36 (0.75) [-0.45 to -0.27] | -0.38 (0.76) [-0.47 to -0.29]
  Sneezing: Change from BL at Week 2 | -0.44 (0.74) [-0.52 to -0.35] | -0.51 (0.69) [-0.59 to -0.42] | -0.40 (0.73) [-0.49 to -0.32]
  Rhinorrhea: Change from BL at Day 3 | -0.37 (0.66) [-0.47 to -0.28] | -0.32 (0.73) [-0.41 to -0.22] | -0.24 (0.74) [-0.33 to -0.15]
  Rhinorrhea: Change from BL at Week 1 | -0.39 (0.77) [-0.49 to -0.29] | -0.38 (0.83) [-0.48 to -0.28] | -0.44 (0.78) [-0.54 to -0.34]
  Rhinorrhea: Change from BL at Week 2 | -0.57 (0.73) [-0.67 to -0.47] | -0.53 (0.83) [-0.63 to -0.43] | -0.56 (0.83) [-0.66 to -0.46]
  Nasal Congestion: Change from BL at Day 3 | -0.22 (0.68) [-0.30 to -0.13] | -0.17 (0.68) [-0.26 to -0.09] | -0.13 (0.65) [-0.22 to -0.04]
  Nasal Congestion: Change from BL at Week 1 | -0.28 (0.81) [-0.38 to -0.18] | -0.22 (0.70) [-0.32 to -0.13] | -0.32 (0.73) [-0.42 to -0.23]
  Nasal Congestion: Change from BL at Week 2 | -0.33 (0.78) [-0.43 to -0.23] | -0.33 (0.75) [-0.43 to -0.23] | -0.37 (0.77) [-0.47 to -0.27]
  Nasal Itching: Change from BL at Day 3 | -0.32 (0.79) [-0.42 to -0.22] | -0.33 (0.82) [-0.43 to -0.23] | -0.15 (0.80) [-0.25 to -0.05]
  Nasal Itching: Change from BL at Week 1 | -0.44 (0.84) [-0.55 to -0.33] | -0.44 (0.88) [-0.55 to -0.34] | -0.35 (0.88) [-0.45 to -0.24]
  Nasal Itching: Change from BL at Week 2 | -0.63 (0.91) [-0.74 to -0.53] | -0.58 (0.86) [-0.68 to -0.48] | -0.52 (0.84) [-0.62 to -0.42]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.547, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.03, 95% CI 2-sided [-0.15 to 0.08] — Difference in LS Means for Change From Baseline in Sneezing Nasal Symptom Sub-Score at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.067, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.10, 95% CI 2-sided [-0.22 to 0.01] — Difference in LS Means for Change From Baseline in Sneezing Nasal Symptom Sub-Score at Week 2
Statistical Analysis 3: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.895, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.01, 95% CI 2-sided [-0.15 to 0.13] — Difference in LS Means for Change From Baseline in Rhinorrhea Nasal Symptom Sub-Score at Week 2
Statistical Analysis 4: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.627, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.03, 95% CI 2-sided [-0.10 to 0.17] — Difference in LS Means for Change From Baseline in Rhinorrhea Nasal Symptom Sub-Score at Week 2
Statistical Analysis 5: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.535, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.04, 95% CI 2-sided [-0.09 to 0.18] — Difference in LS Means for Change From Baseline in Nasal Congestion Nasal Symptom Sub-Score at Week 2
Statistical Analysis 6: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.557, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.04, 95% CI 2-sided [-0.10 to 0.18] — Difference in LS Means for Change From Baseline in Nasal Congestion Nasal Symptom Sub-Score at Week 2
Statistical Analysis 7: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.119, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.11, 95% CI 2-sided [-0.25 to 0.03] — Difference in LS Means for Change From Baseline in Nasal Itching Nasal Symptom Sub-Score at Week 2
Statistical Analysis 8: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.403, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.06, 95% CI 2-sided [-0.20 to 0.08] — Difference in LS Means for Change From Baseline in Nasal Itching Nasal Symptom Sub-Score at Week 2

6. Secondary Outcome: Change From Baseline in Nasal Finding Score Assessed by the Investigator
Description: The investigator conducted rhinoscopic examinations on participants to evaluate: swelling of inferior nasal concha mucosa (INCM) (score of 0=none to 3=middle nasal concha is not visible), coloring of inferior nasal concha mucosa (INCM) (score of 0=normal to 3=pale), and nasal discharge production (NDP) (score of 0=none to 3=congesting). The score for each nasal finding component could range from 0 to 3, with a higher score indicating more severe symptoms.
Time Frame: Baseline and Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for nasal finding score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Swelling of INCM: Change from BL at Day 3 | -0.23 (0.70) [-0.32 to -0.14] | -0.17 (0.68) [-0.26 to -0.08] | -0.13 (0.71) [-0.22 to -0.05]
  Swelling of INCM: Change from BL at Week 1 | -0.35 (0.71) [-0.44 to -0.25] | -0.31 (0.69) [-0.40 to -0.21] | -0.34 (0.78) [-0.43 to -0.24]
  Swelling of INCM: Change from BL at Week 2 | -0.38 (0.74) [-0.48 to -0.28] | -0.34 (0.71) [-0.44 to -0.24] | -0.32 (0.82) [-0.41 to -0.22]
  Coloring of INCM: Change from BL at Day 3 | -0.27 (0.86) [-0.37 to -0.16] | -0.26 (0.79) [-0.36 to -0.15] | -0.26 (0.81) [-0.36 to -0.15]
  Coloring of INCM: Change from BL at Week 1 | -0.35 (0.88) [-0.47 to -0.24] | -0.38 (0.89) [-0.49 to -0.27] | -0.40 (0.91) [-0.51 to -0.28]
  Coloring of INCM: Change from BL at Week 2 | -0.48 (0.97) [-0.60 to -0.36] | -0.48 (0.85) [-0.60 to -0.37] | -0.45 (0.96) [-0.57 to -0.33]
  NDP: Change from BL at Day 3 | -0.23 (0.76) [-0.32 to -0.14] | -0.24 (0.75) [-0.32 to -0.15] | -0.18 (0.65) [-0.27 to -0.09]
  NDP: Change from BL at Week 1 | -0.33 (0.75) [-0.42 to -0.24] | -0.36 (0.75) [-0.45 to -0.26] | -0.41 (0.75) [-0.50 to -0.31]
  NDP: Change from BL at Week 2 | -0.41 (0.71) [-0.51 to -0.32] | -0.38 (0.76) [-0.48 to -0.29] | -0.44 (0.76) [-0.54 to -0.35]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.376, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.06, 95% CI 2-sided [-0.20 to 0.07] — Difference in LS Means for Change From Baseline in Swelling of INCM at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.714, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.03, 95% CI 2-sided [-0.16 to 0.11] — Difference in LS Means for Change From Baseline in Swelling of INCM at Week 2
Statistical Analysis 3: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.725, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.03, 95% CI 2-sided [-0.19 to 0.13] — Difference in LS Means for Change From Baseline in Coloring of INCM at Week 2
Statistical Analysis 4: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.708, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.03, 95% CI 2-sided [-0.19 to 0.13] — Difference in LS Means for Change From Baseline in Coloring of INCM at Week 2
Statistical Analysis 5: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.680, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.03, 95% CI 2-sided [-0.10 to 0.16] — Difference in LS Means for Change From Baseline in NDP at Week 2
Statistical Analysis 6: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.373, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.06, 95% CI 2-sided [-0.07 to 0.19] — Difference in LS Means for Change From Baseline in NDP at Week 2

7. Secondary Outcome: Change From Baseline in Eye Symptom Score Assessed by the Investigator
Description: The investigator interviewed and examined participants for eye (itching) symptoms (score of 0=none to 3=eye is itchy, requiring frequent rubbing of eye). Eye symptom scores could range from 0 to 3, with a higher score indicating greater eye itchiness.
Time Frame: Baseline and Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for eye symptom score as assessed by the investigator.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Change from BL at Day 3 | -0.17 (0.76) [-0.27 to -0.08] | -0.24 (0.71) [-0.34 to -0.15] | -0.13 (0.74) [-0.22 to -0.04]
  Change from BL at Week 1 | -0.28 (0.76) [-0.38 to -0.18] | -0.35 (0.76) [-0.44 to -0.25] | -0.26 (0.83) [-0.36 to -0.16]
  Change from BL at Week 2 | -0.38 (0.84) [-0.48 to -0.28] | -0.44 (0.77) [-0.54 to -0.34] | -0.37 (0.79) [-0.46 to -0.27]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.849, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.01, 95% CI 2-sided [-0.14 to 0.12] — Difference in LS Means for Change From Baseline in Eye Symptom Score at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.260, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.07, 95% CI 2-sided [-0.20 to 0.06] — Difference in LS Means for Change From Baseline in Eye Symptom Score at Week 2

8. Secondary Outcome: Number of Participants With Moderate-to-Remarkable Improvement in Global Improvement Assessed by the Investigator
Description: The investigator comprehensively evaluated participants on global improvement according to 5 grades: 1=remarkably improved, 2= moderately improved, 3=slightly improved, 4=unchanged, and 5=aggravated. The number of participants who were evaluated as remarkably improved and moderately improved was calculated.
Time Frame: Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for global improvement.
Measure: Number; unit: Participants
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 200 | 203 | 201
Participants
  Day 3 (n=199, 201, 200) | 67 | 61 | 53
  Week 1 (n=200, 203, 201) | 72 | 83 | 91
  Week 2 (n=200, 203, 201) | 96 | 93 | 106
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.340, Regression, Logistic; Logistic model with global improvement rate as response variable and treatment, age strata, and severity as factors; Odds Ratio (OR) = 0.826, 95% CI 2-sided [0.558 to 1.223] — Difference in the number of participants with moderate or remarkable improvement at Week 2. An odds ratio >1 is in favor of the first group of the pairwise comparison
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.159, Regression, Logistic; Logistic model with global improvement rate as response variable and treatment, age strata, and severity as factors; Odds Ratio (OR) = 0.755, 95% CI 2-sided [0.510 to 1.116] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Score on Interference With Daily Activities Assessed by the Investigator
Description: The investigator interviewed participants at Baseline, Day 3, Week 1 and Week 2 to evaluate interference with daily activities according to the following scale: 0=none, 1=nasal symptom interferes with daily activities from time to time (+), 2=between 1 and 3 (++), and 3=nasal symtom interferes with daily activity often (+++). Interference with daily activities scores could range from 0 to 3, with a higher score indicating greater interference with daily activities.
Time Frame: Baseline and Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for interference with daily activities.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Change from BL at Day 3 | -0.18 (0.63) [-0.26 to -0.10] | -0.19 (0.58) [-0.27 to -0.12] | -0.07 (0.62) [-0.15 to 0.00]
  Change from BL at Week 1 | -0.22 (0.69) [-0.30 to -0.13] | -0.21 (0.68) [-0.29 to -0.12] | -0.20 (0.64) [-0.28 to -0.11]
  Change from BL at Week 2 | -0.25 (0.73) [-0.34 to -0.16] | -0.29 (0.69) [-0.38 to -0.20] | -0.27 (0.71) [-0.36 to -0.19]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.705, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.02, 95% CI 2-sided [-0.09 to 0.14] — Difference in LS Means for Change from Baseline in Interference with Daily Activities at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.782, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.02, 95% CI 2-sided [-0.13 to 0.10] — Difference in LS Means for Change from Baseline in Interference with Daily Activities at Week 2

10. Secondary Outcome: Change From Baseline in Nasal Symptom Sub-Scores Reported in Participant Diaries
Description: Participants evaluated themselves in their daily allergy diaries for nasal symptoms of: sneezing (daily frequency of attacks; score of 0=less than 1 time to 3=11+ times), rhinorrhea (daily frequency of blowing nose; score of 0=less than 1 time to 3=11+ times), nasal congestion (score of 0=less than nasal blockage without oral breathing to 3=severe nasal blockage causing prolonged oral breathing in a day), and nasal itching (score of 0=none to 3=nose is itchy, requiring frequent rubbing or blowing nose). Each nasal symptom sub-score could range from 0 to 3, with a higher sub-score indicating more frequent/severe nasal symptoms.
Time Frame: Baseline and Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for participant-rated nasal symptom score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Sneezing: Change from BL at Day 3 | -0.27 (0.72) [-0.36 to -0.18] | -0.32 (0.76) [-0.41 to -0.23] | -0.23 (0.79) [-0.32 to -0.13]
  Sneezing: Change from BL at Week 1 | -0.38 (0.72) [-0.48 to -0.29] | -0.40 (0.84) [-0.49 to -0.30] | -0.30 (0.75) [-0.39 to -0.20]
  Sneezing: Change from BL at Week 2 | -0.43 (0.81) [-0.54 to -0.32] | -0.45 (0.86) [-0.55 to -0.35] | -0.33 (0.81) [-0.44 to -0.23]
  Rhinorrhea: Change from BL at Day 3 | -0.20 (0.76) [-0.30 to -0.11] | -0.29 (0.74) [-0.39 to -0.19] | -0.17 (0.80) [-0.27 to -0.08]
  Rhinorrhea: Change from BL at Week 1 | -0.29 (0.81) [-0.39 to -0.18] | -0.36 (0.81) [-0.46 to -0.26] | -0.34 (0.84) [-0.44 to -0.23]
  Rhinorrhea: Change from BL at Week 2 | -0.33 (0.85) [-0.45 to -0.22] | -0.38 (0.86) [-0.50 to -0.27] | -0.45 (0.88) [-0.57 to -0.34]
  Nasal Congestion: Change from BL at Day 3 | -0.18 (0.71) [-0.28 to -0.09] | -0.17 (0.73) [-0.27 to -0.08] | -0.18 (0.75) [-0.28 to -0.09]
  Nasal Congestion: Change from BL at Week 1 | -0.23 (0.69) [-0.33 to -0.13] | -0.24 (0.79) [-0.34 to -0.14] | -0.25 (0.83) [-0.35 to -0.15]
  Nasal Congestion: Change from BL at Week 2 | -0.23 (0.76) [-034 to -0.12] | -0.26 (0.88) [-0.37 to -0.15] | -0.32 (0.78) [-0.43 to -0.20]
  Nasal Itching: Change from BL at Day 3 | -0.29 (0.76) [-0.39 to -0.19] | -0.35 (0.85) [-0.45 to -0.25] | -0.22 (0.77) [-0.33 to -0.12]
  Nasal Itching: Change from BL at Week 1 | -0.40 (0.88) [-0.51 to -0.30] | -0.42 (0.80) [-0.53 to -0.32] | -0.39 (0.87) [-0.50 to -0.29]
  Nasal Itching: Change from BL at Week 2 | -0.52 (0.92) [-0.64 to -0.40] | -0.47 (0.90) [-0.59 to -0.36] | -0.44 (0.87) [-0.56 to -0.33]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.175, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.10, 95% CI 2-sided [-0.24 to 0.04] — Difference in LS Means for Change from Baseline in Sneezing at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.098, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.12, 95% CI 2-sided [-0.26 to 0.02] — Difference in LS Means for Change from Baseline in Sneezing at Week 2
Statistical Analysis 3: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.130, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.12, 95% CI 2-sided [-0.04 to 0.27] — Difference in LS Means for Change from Baseline in Rhinorrhea at Week 2
Statistical Analysis 4: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.375, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.07, 95% CI 2-sided [-0.08 to 0.22] — Difference in LS Means for Change from Baseline in Rhinorrhea at Week 2
Statistical Analysis 5: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.285, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.08, 95% CI 2-sided [-0.07 to 0.24] — Difference in LS Means for Change from Baseline in Nasal Congestion at Week 2
Statistical Analysis 6: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.490, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.05, 95% CI 2-sided [-0.10 to 0.21] — Difference in LS Means for Change from Baseline in Nasal Congestion at Week 2
Statistical Analysis 7: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.345, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.08, 95% CI 2-sided [-0.23 to 0.08] — Difference in LS Means for Change from Baseline in Nasal Itching at Week 2
Statistical Analysis 8: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.699, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.03, 95% CI 2-sided [-0.19 to 0.13] — Difference in LS Means for Change from Baseline in Nasal Itching at Week 2

11. Secondary Outcome: Change From Baseline in Eye Symptom Score Reported in Participant Diaries
Description: Participants evaluated themselves in their daily allergy diaries for eye (itching) symptoms (score of 0=none to 3=eye is itchy, requiring frequent rubbing of eye). Eye symptom scores could range from 0 to 3, with a higher score indicating greater eye itchiness.
Time Frame: Baseline and Day 3, Week 1, Week 2
Population: The FAS population consisted of all participants who took at least one dose of study drug and had a baseline or at least one post-baseline assessment for participant-rated eye symptom score.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Number analyzed (Participants) | 202 | 203 | 201
Score on a Scale
  Change from BL at Day 3 | -0.28 (0.73) [-0.38 to -0.19] | -0.25 (0.72) [-0.34 to -0.15] | -0.20 (0.83) [-0.30 to -0.11]
  Change from BL at Week 1 | -0.31 (0.82) [-0.40 to -0.21] | -0.33 (0.75) [-0.43 to -0.24] | -0.26 (0.80) [-0.35 to -0.16]
  Change from BL at Week 2 | -0.33 (0.80) [-0.44 to -0.22] | -0.35 (0.82) [-0.45 to -0.24] | -0.27 (0.84) [-0.38 to -0.17]
Statistical Analysis 1: Comparison: Desloratadine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.414, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.06, 95% CI 2-sided [-0.20 to 0.08] — Difference in LS Means for Change from Baseline in Eye Symptom Score at Week 2
Statistical Analysis 2: Comparison: Desloratadine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.281, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.08, 95% CI 2-sided [-0.22 to 0.06] — Difference in LS Means for Change from Baseline in Eye Symptom Score at Week 2

ADVERSE EVENTS:
Time Frame: Up to 2 weeks after last dose of study drug (up to 4 weeks)
Description: The population consisted of all participants who received at least one dose of study drug.
Arm/Group | Desloratadine 5 mg | Desloratadine 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/202 | 0/203 | 0/201
Other Adverse Events (participants affected / at risk) | 11/202 | 17/203 | 9/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine 5 mg (N=202) | Desloratadine 10 mg (N=203) | Placebo (N=201)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine 5 mg (N=202) | Desloratadine 10 mg (N=203) | Placebo (N=201)
Nasphopharyngitis (Infections and infestations) | 11 (12) | 17 (17) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.